CLINICAL TRIAL: NCT06423859
Title: A Comparative Study Between Articaine Alone Versus Articaine Plus Dexmedetomidine for Ambulatory Orthopedic Surgery Under Supraclavicular Block
Brief Title: Articaine Plus Dexmedetomidine in Supraclavicular Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Samar Rafik Mohamed Amin, Assistant professor of anaesthesia and intensive care, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC 19-1-2024
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Post Operative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative | interventions — Carticaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Articaine alone (Active Comparator): supraclavicular brachial plexus block will be performed in this group guided by ultrasound. A 30 ml volume local anesthetic will be injected in the form of (29 cc articaine 2% + 1 cc isotonic saline)
  Interventions: Drug: Articaine
- Articaine and Dexmedetomidine (Experimental): supraclavicular brachial plexus block will be performed in this group guided by ultrasound. A 30 ml volume local anesthetic will be injected in the form of (29 cc articaine 2% + 1 cc volume of Dexmedetomidine 1 ug/kg)
  Interventions: Drug: Articaine; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Articaine — supraclavicular brachial plexus block with articaine 2%
Drug: Dexmedetomidine — supraclavicular brachial plexus block with articaine 2% in addition with Dexmedetomidine
  Arms: Articaine and Dexmedetomidine

SUMMARY:
Articaine has emerged as a local anesthetic (LA) that produces sensory and motor blockade shorter than bupivacaine and lower in neurotoxicity than lidocaine.

Studies have shown that adding dexmedetomidine to LA produces prolongation of sensory and motor bock duration.

Early regain of motor power with adequate analgesia is needed in ambulatory surgery, for early start of physiotherapy. This study was designed to test efficacy of adding dexmedetomidine to articaine on the duration of sensory and motor block.

DETAILED DESCRIPTION:
Articaine is an amide LA produced in the 1960s and first used in clinical trials in 1974. Although it is an amide that is similar to prilocaine in chemical structure, it contains a thiophene ring rather than a benzene ring. Articaine is a rapid and short acting LA, which has low neurotoxicity and appears to diffuse through tissues more readily than other commonly used LA agents. It is metabolized by nonspecific plasma esterases both in blood and tissues, leading to its rapid clearance.

α2-adrenergic receptor agonists have been the focus of interest for their sedative, analgesic, perioperative sympatholytic, and cardiovascular stabilizing effects along with providing reduction in anesthetic requirements. Dexmedetomidine may act on supraspinal (locus coeruleus) or spinal level or peripheral α2-adrenoreceptor to reduce nociceptive transmission, leading to analgesia.

Previous trials focused on adding dexmedetomidine to either levobupivacaine and bupivacaine, found augmentation of both sensory and motor block along with prolonged duration of effective analgesia. However, there remains limited knowledge of the analgesic efficacy and clinical utility of adding dexmedetomidine to articaine during peripheral nerve block in humans.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-60 years planned for upper limb surgery below the midhumerus with an expected time of less than 90 min usually under tourniquet.

Exclusion Criteria:

* allergies to local anesthetic,
* those with ASA III and IV,
* patients who refuse to participate,
* uncooperative patients,
* patients who have infection at the site of injection,
* patients who have bleeding disorder, and patients on anticoagulant drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Sensory block duration | 24 hours post block
  the time between the onset of sensory block to the complete resolution of anesthesia on all nerves distribution.

SECONDARY OUTCOMES:
onset time of sensory block | 15 minutes after block
  The time between the end of the drug injection and the total abolition of pinprick sensation along the distribution of any of nerves - median, ulnar, radial, or musculocutaneous
onset time for motor block | 15 minutes after block
  the time between the end of the drug injection and Grade 1 motor block
motor duration block | 24 hours post block
  the time interval between the onset time of motor block and the recovery of complete motor function of that limb
Analgesia time | 24 hours postoperative
  time interval between the administration of local anesthesia solution and onset of pain at surgical site

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Rafik Mohamed Amin, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided